CLINICAL TRIAL: NCT01774513
Title: EUS-guided Procore-biopsy in Diagnosing Autoimmune Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1212013
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Autoimmune Pancreatitis
MeSH Terms: conditions — Autoimmune Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Procore Needle (Experimental)
  Interventions: Device: Procore-Needle

INTERVENTIONS:
Device: Procore-Needle

SUMMARY:
The goal of this prospective study is to evaluate the feasibility of the Core Biopsy Needle with reverse bevel (Procore TM) in diagnosing autoimmune pancretitis

ELIGIBILITY:
Inclusion Criteria:

* patient age 18 years and older
* patients with suspicion of autoimmune pancreatitis (based on the findings in EUS and MRI)

Exclusion Criteria:

* unable to obtain informed consent
* ASA class 4 and 5
* known pregnancy
* contraindication for endoscopy or for biopsy sampling
* patients with high suspicion on pancreatic cancer (based on the findings in radiology and EUS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic yield | 6 months
  Number of patients with adequate tissue sample (which allows definitive diagnosis)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany